CLINICAL TRIAL: NCT02929420
Title: A Multicenter, Randomized, Open, Parallel Controlled Clinical Study on the Efficacy and Safety of the Treatment of Cyclomastopathy With Xiaoru Sanjie Capsule
Brief Title: A Clinical Study on the Efficacy and Safety of the Treatment of Hyperplasia of Mammary Glands With Xiaoru Sanjie Capsule
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ry-2016-08
Record Dates: First submitted 2016-08-23; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Fibrocystic Disease of Breast
Keywords: Multicenter; randomized; open; parallel controlled
MeSH Terms: conditions — Fibrocystic Breast Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xiaoru Sanjie capsules (Experimental): a new recipe of traditional chinese medicine； Xiaoru Sanjie capsules,three pills every time,three time a day,PO, last three months.
  Interventions: Drug: Xiaoru Sanjie capsules
- Xiao Yao pills (Placebo Comparator): a kind of traditional chinese medicine that is efficient and safe to treat hyperplasia of mammary glands.
  Xiaoyao pills,three pills every time,three time a day,PO,last three months.
  Interventions: Drug: Xiao Yao pills

INTERVENTIONS:
Drug: Xiaoru Sanjie capsules — Oral medication for a total of 90 days. According to the instructions, P.O., three times a day, each time three tablets, take a month as a treatment course, continuous use of 3 courses.
  Other Names: Xiaoru Sanjie capsule
  Arms: Xiaoru Sanjie capsules
Drug: Xiao Yao pills — Oral medication for a total of 90 days. According to the instructions, P.O., three times a day, each time three tablets, take a month as a treatment course, continuous use of 3 courses.
  Other Names: ease pills
  Arms: Xiao Yao pills

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Xiaoru Sanjie capsule in the treatment of cyclomastopathy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open and parallel controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old female patients with cyclomastopathy who signed a written informed consent.
* The subjects voluntarily entered the clinical observation whom are hospitalized patients or outpatients with good compliance.
* They have specific symptoms, such as distending pain of the breast, stabbing pain, dull pain and radiating pain.
* They have specific physical sign, for example, we can touch block gland, granular, nodular or cord like glands and etc..
* Breast ultrasound or molybdenum target show I-III class by Breast Imaging Reporting and Data System.

Exclusion Criteria:

* Women who are pregnant or lactating, and who has the history of periarthritis of shoulder.
* Excluding breast fibrocellular tumor, breast cancer and other breast diseases.
* Patients with poor self coordination, mentally retarded patients, or have cardiovascular and cerebrovascular disease, severe organic disease, as well as the hematopoietic system disease or mental illness.
* Be judged as over middle degree depression by the Hamilton's depression scale.
* Allergic constitution patients, and people who are allergic to a variety of drugs.
* Any medical history which may interfere with the test results or increase the risk of patients according to the investigators.
* Patients who have received treatment of other diseases, and those treatment methods and targets may have an impact on the indicators of this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the size of breast lumps | after 30 days' treatment
  Assess the size of breast lumps by breast ultrasonography or breast molybdenum target.
the size of breast lumps | after 60 days' treatment
  Assess the size of breast lumps by breast ultrasonography or breast molybdenum target.
the size of breast lumps | after 90 days' treatment
  Assess the size of breast lumps by breast ultrasonography or breast molybdenum target.
the scope of breast lumps | after 30 days' treatment
  Assess the scope of breast lumps by breast ultrasonography or breast molybdenum target.
the scope of breast lumps | after 60 days' treatment
  Assess the scope of breast lumps by breast ultrasonography or breast molybdenum target.
the scope of breast lumps | after 90 days' treatment
  Assess the scope of breast lumps by breast ultrasonography or breast molybdenum target.
the hardness of breast lumps | after 30 days' treatment
  Assess the hardness of breast lumps by breast ultrasonography or breast molybdenum target.
the hardness of breast lumps | after 60 days' treatment
  Assess the hardness of breast lumps by breast ultrasonography or breast molybdenum target.
the hardness of breast lumps | after 90 days' treatment
  Assess the hardness of breast lumps by breast ultrasonography or breast molybdenum target.
pain of breast | after 30 days' treatment
  According to hyperplasia of mammary glands efficacy appraisal standard of 2002 china association of chinese medicine surgery branch.
pain of breast | after 60 days' treatment
  According to hyperplasia of mammary glands efficacy appraisal standard of 2002 china association of chinese medicine surgery branch.
pain of breast | after 90 days' treatment
  According to hyperplasia of mammary glands efficacy appraisal standard of 2002 china association of chinese medicine surgery branch.

SECONDARY OUTCOMES:
all adverse reactions after taking Xiaoru Sanjie capsule | after 30 days' treatment
  Number of Participants with different adverse reactions after taking treatment.
all adverse reactions after taking Xiaoru Sanjie capsule | after 60 days' treatment
  Number of Participants with different adverse reactions after taking treatment.
all adverse reactions after taking Xiaoru Sanjie capsule | after 90 days' treatment
  Number of Participants with different adverse reactions after taking treatment.
the level of estrogen | after 30 days' treatment
the level of estrogen | after 60 days' treatment
the level of estrogen | after 90 days' treatment
the level of progestin | after 30 days' treatment
the level of progestin | after 60 days' treatment
the level of progestin | after 90 days' treatment
the level of prolactin | after 30 days' treatment
the level of prolactin | after 60 days' treatment
the level of prolactin | after 90 days' treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yu Ren, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Yu Ren, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes